CLINICAL TRIAL: NCT00548353
Title: A Randomized, Double-Blind, Placebo Controlled, 2-Period, Fixed-Sequence Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profile of Orally Administered MK3207 in Patients During and Between Their Acute Migraine Attacks
Brief Title: A Study of Gastric Delay in Migraine Patients (3207-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3207-003; MK3207-003; 2007_599
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — 2-(8-(3,5-difluorophenyl)-10-oxo-6,9-diazaspiro(4.5)dec-9-yl)-N-(2'-oxo-1,1',2',3-tetrahydrospiro(indene-2,3'-pyrrolo(2,3-b)pyridin)-5-yl)acetamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): MK3207 Orally administered to patients with water. During each period (with and without acute migraine).
  Interventions: Drug: MK3207
- 2 (Placebo Comparator): MK3207 placebo as tablets will be Orally administered to patients with water. During each period (with and without acute migraine).
  Interventions: Drug: Comparator: Placebo (unspecified)

INTERVENTIONS:
Drug: MK3207 — M3207 (20 mg); patients will be administered a single dose of 100 mg of MK3207 (i.e., 5 x20-mg tablets).
  Arms: 1
Drug: Comparator: Placebo (unspecified) — M3207 (20 mg) Pbo; patients will be administered a single dose of 100 mg of MK3207 Pbo (i.e., 5 x20-mg tablets).
  Arms: 2

SUMMARY:
A study to assess safety and PK of an investigational drug in migraine patients during and between migraine attacks.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking male or female between 18 to 45 years of age
* Patient typically has between 2 and 10 migraine attacks per month, rated as moderate or severe

Exclusion Criteria:

* Patient has any other medical conditions other than migraine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Safety in migraine patients | 12 Weeks

SECONDARY OUTCOMES:
PK in migraine patients | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC